CLINICAL TRIAL: NCT05960357
Title: State Anxiety Levels of Pregnant Women Who Were Given or Not Given Information About the Fetus With Ultrasound Images During Detailed Ultrasound: A Randomized Controlled Study
Brief Title: State Anxiety Levels of Pregnant Women to Inform About Fetus With Ultrasound Images During Detailed Ultrasound.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Özlem KOÇ, assistant professor, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: aybars2019
Record Dates: First submitted 2023-07-14; First posted 2023-07-25 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2023-07

CONDITIONS: Ultrasound; Perinatal Care; Anxiety
Keywords: Ultrasound; Perinatal care; To inform; Consultancy; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Informed group during Ultrasound Examination (Experimental): Before starting the detailed USG examination for the experimental group, Personal Information Form and State-Anxiety Inventory will be filled. While informing about the fetus during the USG examination, the pregnant woman will be informed by using the physical images of the fetus (hand, arm, face, heartbeat, information about the internal organs, etc.) using the USG screen. After the USG is completed, the State-Anxiety Inventory will be filled again as a final test.
  Interventions: Other: To inform
- Control group (No Intervention): In the control group, the Personal Information Form and the State-Anxiety Inventory will be filled before the USG procedure, and only the State-Anxiety Inventory after the USG procedure. After the data collection process is completed, the pregnant woman will be informed about the USG results.

INTERVENTIONS:
Other: To inform — It includes providing all necessary information about the fetus to the pregnant woman by using the ultrasound monitor during the detailed ultrasound.
  Arms: Informed group during Ultrasound Examination

SUMMARY:
The aim of the study is to determine the state anxiety levels of the pregnant women who were given and not given information about the fetus with USG images during the detailed ultrasound (USG) and to compare them in both groups. This research is in the design of pre-test-post-test applied and randomized controlled research. Dependent variables: State anxiety levels Independent variables: Being informed during ultrasound Control variables: Socio-demographic variables and obstetric variables.

DETAILED DESCRIPTION:
The research population will be composed of pregnant women who applied to the perinatology polyclinic of the Fırat University Hospital, Department of Obstetrics and Gynecology for detailed USG. The sample size was calculated using the G*Power V. 3.1.9.7 program. According to the results of 95% confidence (1-α), 95% test power (1-β), d=0.72 effect size and two-way independent samples t test power analysis, 51 in each group, a total of at least 102 people were sampled. was calculated (Ekrami et al., 2019).

Randomization

Pregnant women who are suitable for the sample selection criteria, using the Random Integer Generator method under Numbers sub-title from Random.org, for the numbers distributed in 2 columns consisting of 1-102 numbers.

Which column would be the experiment and which column would be the control was determined by drawing lots.

Pre-test-Post-test application

Before starting the detailed USG examination for the experimental group, Personal Information Form and State-Anxiety Inventory (DCI) will be filled. While informing about the fetus during the USG examination, the pregnant woman will be informed by using the physical images of the fetus (hand, arm, face, heartbeat, information about the internal organs, etc.) using the USG screen. After the USG is completed, the State-Anxiety Inventory (DCI) will be filled again as a final test. In the control group, the Personal Information Form and State-Anxiety Inventory (DCI) will be filled before the USG procedure, and only the State-Anxiety Inventory (DCI) after the USG procedure. After the data collection process is completed, the pregnant woman will be informed about the USG results.

ELIGIBILITY:
Inclusion Criteria:

* 18-23. in gestational week
* Not carrying any risk factors (pre-eclampsia, IUGG, premature rupture of membranes, getational diabetes, etc.) during pregnancy,
* Pregnant women who did not have any diagnosed problems related to the health of the fetus (such as fetal anomaly, intrauterine growth retardation) were included in the study.

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Personal Information Form | through study completion, an average of 1 year
  The Personal Information Form developed by the researchers consists of questions that determine some descriptive characteristics of pregnant women. (age, education level, employment status, income status, number of living children, number of pregnancies, current gestational week).

SECONDARY OUTCOMES:
State-Anxiety Inventory | through study completion, an average of 1 year
  The Turkish validity and reliability study of the inventory developed by Spielberger et al. was performed by Öner and Le Compte (1983), and the Cronbach's alpha coefficient was found to be 0.83 (Öner & LeCompte, 1985). The 20-item scale consists of items describing how people feel under certain conditions at a certain time and their feelings about the situation they are in (For example, 'I am calm at the moment'). The scale consists of 4-point Likert-type responses as (1) not at all, (2) a little, (3) a lot, (4) completely. There are ten (items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20) reversed statements in the scale. The score obtained from the scale varies between 20 and 80. High scores on the scale indicate high anxiety, low scores indicate mild anxiety (Öner & LeCompte, 1985).

CONTACTS AND LOCATIONS:
Locations (1):
- Tarsus University, Mersin, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No